CLINICAL TRIAL: NCT05059678
Title: Parenting Support Intervention for Families Coping With an Advanced Cancer Diagnosis
Brief Title: Parenting Support Intervention for Families Coping With Metastatic or Locally Recurrent Solid Tumor Diagnosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-0380; NCI-2021-09153 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0380 (Other: M D Anderson Cancer Center); R21CA256694 (NIH)
Record Dates: First submitted 2021-09-10; First posted 2021-09-28 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Malignant Solid Neoplasm; Recurrent Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Practice Guidelines as Topic; Standard of Care; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (education material, videoconference session) (Experimental): Examine the acceptability of a parenting support intervention in 10 patients with an incurable cancer and their spousal caregivers (cohort A) and 10 patients with an advanced cancer diagnosis and their family caregivers (cohort B).
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration
- Group II (waitlist control) (Active Comparator): Participants receive standard of care.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
  Arms: Group II (waitlist control)
Other: Educational Intervention — Receive educational materials and attend videoconference sessions
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group I (education material, videoconference session)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial examines the acceptability and effect of a parenting support intervention for families coping with solid tumor that has spread to other places in the body (metastatic) or has come back (recurrent). Parenting support program may help to reduce common parenting concerns, improve communication between parents and children about cancer, and improve the overall psychological wellbeing of parents.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine the acceptability a parenting support intervention in 10 patients with an incurable cancer and their spousal caregivers. (Trial 1) II. Examine the feasibility of implementing a parenting support intervention in 50 patients with an incurable cancer and their spousal caregivers. (Trial 2) III. Evaluate the initial evidence for intervention efficacy relative to waitlist control (WLC) group regarding patient and spousal caregiver psychological symptoms (primary outcome) and parenting concerns and parenting efficacy (secondary outcomes) and patient end of life (EOL) healthcare utilization (exploratory outcome). (Trial 2) IV. Understand the patients and caregivers' experiences using qualitative methods regarding participation in this study and explore emerging themes as possible intervention mediators/moderators to be examined in future research. (Trial 2)

OUTLINE:

TRIAL 1: Participants receive education materials (brochure and a video) and attend 2 weekly videoconference intervention sessions over 45 minutes each. Caregivers attend 2 additional weekly intervention sessions over 45 minutes each.

TRIAL 2: Participants are randomized to 1 of 2 groups.

GROUP I: Participants receive education materials (brochure and a video) and attend 2 weekly videoconference intervention sessions over 45 minutes each. Caregivers attend 2 additional weekly intervention sessions over 45 minutes each.

GROUP II: Participants receive standard of care.

After completion of study, participants in Trial 1 are followed up at 6 and 12 weeks and participants in Trial 2 are followed up at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants must (1) be diagnosed with a metastatic or locally recurrent solid malignant tumor and on active treatment; (2) be at least 18 years old; (3) have at least one dependent child between the ages of 4 and 16 and currently living with the parent; (4) be able to provide informed consent and (5) have a spousal caregiver over the age of 18 who co-parents the child(ren) (i.e. share custody) and is willing and able to consent to participate.*

Exclusion Criteria:

* Participants and caregivers who do not read and speak English and who do not have access to the internet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Examine the feasibility of implementing a parenting support intervention in 50 patients with an incurable cancer and their spousal caregivers. | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Milbury, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center — http://www.mdanderson.org